CLINICAL TRIAL: NCT04643444
Title: Police Officer COVID-19 Seroprevalence Survey in the Canton of Bern, Switzerland
Brief Title: Police COVID-19 Serosurvey
Acronym: PoliCOV
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Interregionale Blutspende SRK Bern (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-02650
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2 Infection; Volunteers; Healthy
Keywords: COVID-19; SARS-COV-2; Antibodies; Seroprevalence
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sampling — Testing for the presence of SARS-CoV-2 antibodies
Other: Online Questionnaire — Questions on working place, risk profiles and PPE

SUMMARY:
The investigators aim to determine the immune status of the employees of the cantonal police of Bern against SARS-CoV-2 over a period of 1 year, and to investigate the risk profile of the study participants and their risk of SARS-CoV-2 exposure in their working and private environments, as well as to evaluate the use of personal protective equipment at potential exposure instances.

DETAILED DESCRIPTION:
i) To determine the extent of infection with seroprevalence data in the special population of police officers of the canton Bern.

ii) To determine risk factors for infection by comparing the proportion of seropositivity (infected versus noninfected individuals). The investigators hypothesize that police officers with fieldwork activity will have a higher seroprevalence than will office and administration personnel. The investigators hypothesize that working in the city of Bern will be associated with a higher seroprevalence than will working in other geographic areas of the canton (i.e. rural area).

iii) To monitor COVID-19 antibody titres and neutralizing capacity over time and to associate them with reinfection rates and infection-free intervals in police officers after accidental contact with a proven COVID-19 case. The investigators hypothesize that in seropositive individuals, there will be a decreasing dynamic of antibody titres over the one-year study period, and hence, a decrease of neutralizing capacity.

ELIGIBILITY:
Inclusion Criteria:

* Police officers of the cantonal police of Bern volunteering to participate in the study.

Exclusion Criteria:

* Refusal or inability to give informed consent or contraindication to venepuncture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees of the cantonal police of Bern, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Seroprevalence | One year
  The variable of primary interest is COVID-19 seropositivity. This variable is measured at five time points over the one-year study period. The following baseline factors may have an influence on the primary endpoint and will be obtained: (i) pre-existing comorbidities, (ii) rural versus city distribution of working place, and (iii) office work versus field work.

SECONDARY OUTCOMES:
Risk profile assessment | One year
  The investigators will assess the proportion of symptomatic and asymptomatic cases among seropositive participants. The investigators will calculate the attack rate in different subgroup. These include (i) study participants with health-related risk factors (age>50 and age>60 years, diabetes, arterial hypertension, cardiovascular disease, chronic pulmonary disease, immune-compromised status due to host diseases, medical treatment, cancer, obesity), (ii) activity-related subgroups (i.e. fieldwork vs office activity), (iii) geography-related subgroups (i.e. city vs rural areas). In follow-up visits, the antibody titers (i.e. dynamic) and the neutralization capacity will be assessed. Thereby, the investigators will determine the change in serum levels of SARS-CoV-2 antibodies over time in seropositive participants.

CONTACTS AND LOCATIONS:
Overall Officials: Parham Sendi, MD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Institute for Infectious Diseases, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sendi P, Baldan R, Thierstein M, Widmer N, Gowland P, Gahl B, Buchi AE, Guntensperger D, Wider M, Blum MR, Tinguely C, Maillat C, Theel ES, Berbari E, Dijkman R, Niederhauser C. A Multidimensional Cross-Sectional Analysis of Coronavirus Disease 2019 Seroprevalence Among a Police Officer Cohort: The PoliCOV-19 Study. Open Forum Infect Dis. 2021 Oct 16;8(12):ofab524. doi: 10.1093/ofid/ofab524. eCollection 2021 Dec. PMID 34888394

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04643444/Prot_SAP_001.pdf